CLINICAL TRIAL: NCT06205342
Title: STEMCAP-1: Safety and Efficacy of Mesenchymal Stem Cells Associated With Chronic Pancreatitis Pain
Brief Title: Safety and Efficacy of Mesenchymal Stem Cells Associated With Chronic Pancreatitis Pain
Acronym: STEMCAP-1
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Hongjun Wang, Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO 00132905; 1UG3DK136705-01 (NIH)
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Chronic Pancreatitis; Chronic Pain
MeSH Terms: conditions — Pancreatitis, Chronic; Chronic Pain

STUDY DESIGN:
Intervention Model Description: This is a pilot, randomized, double-blind, placebo-controlled, stratified randomization study to determine the efficacy of a single intravenous infusion of allogeneic bone marrow-derived mesenchymal stromal cells in subjects with painful chronic pancreatitis (CP).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Cohort (Experimental): MSC
  Interventions: Drug: Mesenchymal Stem Cells
- Validation Cohort (Placebo Comparator): Placebo
  Interventions: Other: Other: Placebo

INTERVENTIONS:
Drug: Mesenchymal Stem Cells — Autologous bone marrow derived MSCs
  Other Names: MSCs
  Arms: Experimental Cohort
Other: Other: Placebo — Control
  Other Names: Controls
  Arms: Validation Cohort

SUMMARY:
This protocol aims to test whether an infusion of allogeneic bone marrow-derived mesenchymal stromal cells (BM-MSCs) can reduce pain associated with chronic pancreatitis (CP) and explore potential mechanisms of MSC action.

DETAILED DESCRIPTION:
Chronic pancreatitis (CP) and chronic pain: CP is a debilitating disease characterized by persistent pancreatic inflammation, irreversible morphological changes (fibrosis) in the pancreas and severe chronic pain. A progressive loss of exocrine and endocrine function occurs during disease progression. The incidence of CP ranges from 1.6 to 23 cases per 100,000 populations per year worldwide and is likely under diagnosed in the general population. CP in the United States results in more than 122,000 outpatient visits and more than 56,000 hospitalizations per year. The poorly understood pathophysiology of CP makes the identification of means to treat the underlying cellular disorder problematic. Abdominal pain has been reported in at least 80-94% of patients. The pain suffered by CP patients is among the worst encountered in medicine, which often leads to opioid addiction. Many CP patients require hospital admission at some stage in their illness. The cause of pain is complex and is mostly unknown. The pathophysiology in pain due to CP is multifactorial, including peripheral nociception, peripheral/pancreatic neuropathy, and neuroplasticity. Achieving satisfactory pain relief remains a challenge. Current management strategies have used a step-up approach in pain medications that often lead to opioid dependence. Among all patients, 40-75% patients will eventually require surgery, after which only 34-52% attain pain relief after pancreas resection. CP pain provides a useful model for the understanding of the mechanisms and treatment of pain syndromes with an identifiable nociceptive source in general as approximately 50 million U.S. adults are suffering from pain. Improving the management of CP pain may translate to other disease states with pain and opioid addiction.

Mesenchymal stromal cells (MSCs) are adult stem cells that can be harvested and expanded for therapy. MSC therapy is an investigational intervention for CP. There is increasing evidence that MSC therapy can effectively target several injury pathways in a variety of fibroinflammatory diseases and can reduce pain while suppressing inflammation, something that most pharmacological interventions cannot accomplish. Data from animal models and clinical trials support the outstanding and durable effects of MSC infusion in the suppression of chronic neurological pain and inflammation associated with knee osteoarthritis, critical limb ischemia, neuropathy, diabetic neuropathy, and others. MSCs migrate to the spinal cord and pre-frontal cortex of neuropathic mice after injection and exert pain relief. A recent study demonstrated that infusion of human MSCs significantly reduced pain, improved pancreatic volume, and reduced fibrosis in CP rodent models.

Rationale of the study: Because MSCs are a novel therapy that may improve chronic pancreatitis pain in animal models and improve chronic pain in other human disease states, these cells are worthy of study. This pilot study will give participants MSCs or placebo for CP subjects with pain. This study will inform future study designs and may lead to MSCs as a standard of care if they are safe and effective.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years old, male or female
2. Definite chronic pancreatitis
3. Patients who are diagnosed with painful CP for more than 6 months may be constant or may have been waxing and waning/remitting.
4. Baseline Izbicki pain score > 30
5. Stable dose of opioids for the past 30 days

Exclusion Criteria:

1. Acute pancreatitis per 2012 revised Atlanta criteria within the last 30 days.

   * The revised Atlanta classification requires that two or more of the following criteria be met for the diagnosis of acute pancreatitis: (a) abdominal pain suggestive of pancreatitis, (b) serum amylase or lipase level greater than three times the upper normal value, or (c) characteristic imaging findings.
2. Chronic pain syndromes other than pancreatitis that require daily use of opioids in the past 30 days.
3. Severe organ failure(s) likely to interfere with clinical pain outcomes within 6 months.
4. HbA1c >10%
5. Laboratory values of WBC <2.0 cells/10^3, Hemoglobin <8 gm/dl, and platelets <100K cells/10^3, AST or ALT > 3 times the upper limit of normal, or creatinine >2.0 mg/dl
6. New York Heart Association Class 2 or higher congestive heart failure
7. Current lung, hematologic, or solid organ malignancy other than skin, or cervical stage 1 cancers within the past 3 years.
8. Subjects with current infection with hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) infection.
9. Active malignancy with the exception of non-melanoma skin cancer.
10. Any subject who has received an investigational drug or device within 30 days before randomization or who is expected to receive an investigational drug or device during this study.
11. Patients with planned endoscopic or surgical intervention, surgical resection or needle drainage of pancreatic structures in the next 6 months.
12. Patients who have had a pancreatic surgery, endoscopic procedure with therapy, or hospitalization related to pancreatitis within the last 90 days
13. Subjects who have had any ongoing alcohol abuse and/or any illegal drug abuse within the past 6 months.
14. Subjects with infected pancreatic pseudocysts or pancreatic walled-off necrotic areas at the time of consent
15. Females who are pregnant or women of childbearing potential (WOCBP) and males with female partners of childbearing potential who are not willing to use adequate contraception during the study
16. Breastfeeding females
17. Subject unwilling to follow the protocol and assessments

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Izbicki pain score (M6 vs. Baseline) | 6 months
  Change in pain as measured by Izbicki pain scores, a validated score for pain in chronic pancreatitis, consist of 4 questions, with a range of 0 (no pain) to 100 (severe, debilitating pain).

SECONDARY OUTCOMES:
Change in pancreatic volume measured by blinded scoring of MRI | Screening, 6 month
  Pancreas volume change
Change in opioid use as measured in average daily morphine equivalents. | Screening, 1 month, 3 month, 6 month
  Average Daily morphine Equivalent
Changes in quality of life | Screening, 1 month, 3 month, 6 month
  Quality of life to be measured by Promise-29-v 2.1 (with generated T-score for each domain)
Change in M-Manheim Severity Index absolute score | Screening, 1 month, 3 month, 6 month
  Severity of Index absolute scores (with lowest severity 0 and highest severity 24 points)

CONTACTS AND LOCATIONS:
Overall Officials: Hongjun Wang, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No